CLINICAL TRIAL: NCT04240236
Title: Effect of Scalp Blocks on Postoperative Nausea & Vomiting & Recovery Profiles After Craniotomy: A Randomized, Double-Blind, and Controlled Study
Brief Title: Scalp Blocks Effect on Postoperative Nausea & Vomiting After Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Raham Hasan Mostafa, MD, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R 54/2019
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Group S received scalp block with 20 ml of 0.5% bupivacaine
  Interventions: Procedure: Scalp block
- Group C (Placebo Comparator): Group C will not have any intervention
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: Scalp block — Patients will be randomly divided into two groups using a computer generated random number chart. Group S received scalp block with 20 ml of 0.5% bupivacaine, whereas Group C will not receive any intervention and will be considered as control group.
  Arms: Group S
Other: Control Group — Patients will be randomly divided into two groups using a computer generated random number chart. Group S received scalp block with 20 ml of 0.5% bupivacaine, whereas Group C will not receive any intervention and will be considered as control group.
  Arms: Group C

SUMMARY:
In this study, the investigators hypothesize that preemptive scalp block in neurosurgical patients may decrease incidence of PONV after craniotomy through decreasing intraoperative inhalational agents' concentration and decreasing intraoperative opioids requirements, with better intraoperative hemodynamics and lesser recovery time

DETAILED DESCRIPTION:
Patients will be recruited after admission to the hospital for surgery. Randomization will be performed using computer-generated random number tables in opaque sealed envelopes prepared by an anesthesiologist who will be not part of the study

Patients will be randomly divided into two groups using a computer generated random number chart. Group S received scalp block with 20 ml of 0.5% bupivacaine, whereas Group C received scalp block using 20 mL normal saline and will be considered as control group.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients,
* aged 18 to 50 years,
* 70-80 kg,
* undergoing elective supratentorial craniotomy

Exclusion Criteria:

* patients under 18 years of age,
* pregnancy,
* emergency surgery,
* patients with a Glasgow Coma Score (GCS) less than 15,
* those with documented allergy to bupivacaine,
* regular communication not possible,
* Patients requiring prolonged mechanical ventilation (> 2 hours after end of surgery) will be also excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
PONV incidence & severity during the 1st 24 hours in ICU. | 24 hours
  The intensity of the PONV was classified as: 0: without PONV, 1: nausea, 2: vomiting and 3: vomiting more than 2 times [8]. In addition, the incidence of PONV, the first time there was need for ondansetron and its total dose was recorded. With PONV score ≥ 2, the investigators used 4 mg ondansetron IV for antiemetic regimen. The total dose over 24 hours (given as divided doses) must not exceed adult dose of 32 mg.

SECONDARY OUTCOMES:
Intraoperative Mean blood pressure in mmHg | 6 hours
  Mean blood pressure will be measured at specific timing coded as follows: Tzero: mean blood pressure will be measured preoperatively as baseline T1: mean blood pressure will be measured after intubation T2: mean blood pressure will be measured after scalp block T3: mean blood pressure will be measured during pinning T4: mean blood pressure will be measured at skin incision Then mean blood pressure will be measured every 15 min for 1 hour, and every 1 hour till end of surgery T-end: mean blood pressure will be measured at skin closure
Total intraoperative fentanyl consumption in microgram | 6 hours
  The bolus dose given at skin incision was not included
Recovery time in minutes | 10 minutes
  It is the time interval between discontinuation of isoflurane and extubation
Intraoperative Heart rate as number of beats per minute | 6 hours
  Heart rate will be measured at specific timing coded as follows: Tzero: Heart rate will be measured preoperatively as baseline T1: Heart rate will be measured after intubation T2: Heart rate will be measured after scalp block T3: Heart rate will be measured during pinning T4: Heart rate will be measured at skin incision Then Heart rate will be measured every 15 min for 1 hour, and every 1 hour till end of surgery T-end: Heart rate will be measured at skin closure

CONTACTS AND LOCATIONS:
Overall Officials: Raham Hasan Mostafa, MD, Principal Investigator — Assistant Lecturer of Anesthesia, Ain Shams University
Locations (1):
- Raham Hasan, Cairo, Egypt